CLINICAL TRIAL: NCT03960671
Title: Therapeutic Drug Monitoring of Anxiolytics in Children
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Wei Zhao (Other)
Responsible Party: Sponsor-Investigator, Wei Zhao, Professor; Head of department of clinical pharmacy and pharmacology, Shandong University
Organization: Shandong University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2019-anxiolytics-001
Record Dates: First submitted 2019-04-27; First posted 2019-05-23 (Actual); Last update posted 2019-05-23 (Actual); Status verified 2019-05

CONDITIONS: Anxiolytics
MeSH Terms: interventions — Midazolam

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Anxiolytics (Experimental): Pediatric patients treated with sedation using anxiolytics
  Interventions: Drug: Midazolam/diazepam/propofol

INTERVENTIONS:
Drug: Midazolam/diazepam/propofol — Therapeutic drug monitoring of anxiolytics

SUMMARY:
In this study, the therapeutic drug monitoring of anxiolytics is carried out among children to obtain the drug concentration, clinical efficacy and safety data of children patients in different gender and age groups. Then the investigators analyze the relationship between blood drug concentration and efficacy and safety, and provide recommendations for the treatment window of anxiolytics in Chinese children.

ELIGIBILITY:
Inclusion Criteria:

* Anxiolytics was used for therapeutic purposes;
* Age:≤18 years;
* Patients with therapeutic concentration monitoring of anxiolytics.

Exclusion Criteria:

* Patients without therapeutic concentration monitoring of anxiolytics;
* The blood concentrations of the patient was not approved by the quality control center
* Use foods or products that inhibit or induce CYP 3A activity.

Ages: 29 Days to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 500 (Estimated)
Dates: Start 2018-08-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Plasma drug concentration | Through study completion, an average of 14 days
  To detect the plasma concentrations of teicoplanin at therapeutic drug monitoring (TDM).

CONTACTS AND LOCATIONS:
Locations (1):
- Shandong Provincial Qianfoshan Hospital, Ji'nan, Shandong, China

IPD SHARING:
Plan to Share IPD: No